CLINICAL TRIAL: NCT05786599
Title: Methadone to Treat Painful Chemotherapy Induced Peripheral Neuropathy (METACIN): a Randomized Double-blind Controlled Trial
Brief Title: Methadone to Treat Painful Chemotherapy Induced Peripheral Neuropathy
Acronym: METACIN
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Mathieos Belayneh, Clinician Researcher, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H22-01702
Record Dates: First submitted 2023-03-09; First posted 2023-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Methadone; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- methadone (Experimental): Methadone is a strong opioid that is μ-opioid receptor agonist like other opioids; however, it is additionally a N-methyl-D- aspartate antagonist with serotonin and norepinephrine reuptake inhibition; these attributes enable its efficacy in neuropathic pain and may prevent opioid tolerance over time. It is commonly used to treat opioid use disorder, as well as to treat severe pain. This medication is taken orally every 8 hours when used to treat pain. It has not been studied to treat chemotherapy-induced peripheral neuropathy.
  Interventions: Drug: methadone
- duloxetine (Active Comparator): Duloxetine is a serotonin and norepinephrine reuptake inhibitor that is commonly used to treat major depressive disorder, generalized anxiety disorder, and neuropathic pain. This medication is taken orally once daily for all of its indications. It is the only well-studied medication that is recommended internationally to treat chemotherapy-induced peripheral neuropathy.
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: methadone — The treatment arm will take methadone 2 mg PO q8h and a placebo called "placeboD" PO qdaily. PlaceboD and duloxetine will be placed in capsules to be virtually indistinguishable.
  Participants will be followed (televisit or in-person) by assessors every week; this will take approximately 15 minutes. This includes review of questionnaire(s), adverse events (and any potential management), and recommendations on dose titration. To maintain blinding and ensure standardization across assessors, titration protocols will be provided. If pain is not controlled, the assessors will instruct the participant to increase their methadone/placeboM drug by 1 capsule PO q8h and their duloxetine/placeboD drug to 2 capsules PO qdaily (the study maximum). If there are poorly tolerated adverse events the dose will be reduced to the previously tolerated dose, and then the following week they may attempt to titrate up again per the above protocol.
  Other Names: metadol
  Arms: methadone
Drug: duloxetine — The control arm will receive duloxetine 30 mg PO qdaily, and a placebo called "placeboM" PO q8h. PlaceboM and methadone will be placed in capsules to be virtually indistinguishable.
  Participants will be followed (televisit or in-person) by assessors every week; this will take approximately 15 minutes. This includes review of questionnaire(s), adverse events (and any potential management), and recommendations on dose titration. To maintain blinding and ensure standardization across assessors, titration protocols will be provided. If pain is not controlled, the assessors will instruct the participant to increase their methadone/placeboM drug by 1 capsule PO q8h and their duloxetine/placeboD drug to 2 capsules PO qdaily (the study maximum). If there are poorly tolerated adverse events the dose will be reduced to the previously tolerated dose, and then the following week they may attempt to titrate up again per the above protocol.
  Other Names: cymbalta
  Arms: duloxetine

SUMMARY:
Chemotherapy induced peripheral neuropathy (CIPN) or nerve pain, is a painful and debilitating complication which can chronically affect up to 70% of patients who receive chemotherapy. It causes "glove-and-stocking" distribution of nerve-pain, weakness, and other debilitating symptoms. This can affect patient's quality of life, function, ability to tolerate chemotherapy, and return to work.

Duloxetine is the only recommended medication to reduce the painful symptoms and consequences of CIPN by national and international groups such as the American Society of Clinical Oncology. However, studies indicate it only has modest effect; for example, the largest study shows it only reduces pain by 0.73/10 points compared to placebo.

Another promising medication in theory and practice is methadone. It is a commonly used and well-studied opioid with unique attributes which allows it to treat non-cancer and cancer associated nerve-pain with better efficacy when compared to other opioids. Furthermore, patients appear to develop less tolerance to methadone over time when compared to other opioids; this is helpful as many develop long-term CIPN and may greatly benefit from long-term pain medication. Therefore, if a patient requires chronic opioids to reduce the painful symptoms of CIPN, one that develops less tolerance is invaluable. Despite the promising role for methadone to treat CIPN, it has not been studied to treat this condition. Therefore, methadone may never be considered by prescribers to reduce the painful symptoms of CIPN.

This study is a randomized controlled trial to assess the efficacy of methadone compared to duloxetine to treat painful CIPN. Participants will be randomized to receive either methadone or duloxetine regularly for 5 weeks. Methadone and duloxetine will be placed in indistinguishable capsules, so the participant and assessor are not aware of their treatment. They will be followed virtually or in-person weekly for 5 weeks where they will answer brief questionnaires detailing the effect of their treatment on their pain and their dose will increase weekly as tolerated until their pain is controlled or its the end of the study. This study would be critical in assessing the efficacy of a very promising medication to reduce the painful symptoms of CIPN: a debilitating disorder with otherwise few treatment options.

DETAILED DESCRIPTION:
Rationale: Chemotherapy-induced peripheral neuropathy (CIPN) is a debilitating consequence of chemotherapy that causes chronic neuropathic pain in up to 70% of cancer patients. Duloxetine is the only pharmacotherapy recommended by international guidelines, and its effects are modest. Methadone is increasingly used to treat refractory neuropathic pain in cancer patients and has not been studied in CIPN.

Question: Is methadone more effective than duloxetine for the treatment of CIPN? Participants: Adult cancer patients with life expectancy greater than 12 weeks who have greater than grade 1 CIPN based on National Cancer Institute Common Toxicity Criteria for Adverse Events version 5.0 grading scale lasting ≥3 months beyond chemotherapy completion.

Intervention: This trial will follow a double-blind double-dummy randomized controlled trial design where participants will be randomized to either treatment arm (methadone) or control arm (duloxetine). They will be followed weekly over a 5-week period and undergo dose titration.

Outcomes: The primary outcome will be efficacy of methadone compared to duloxetine to reduce the average pain intensity between the baseline and end of study for patients with painful CIPN. Secondary outcomes include i) Determine the effect of methadone compared to duloxetine to improve functional interference using the Brief Pain Inventory-Short Form; ii) Determine the effect of methadone compared to duloxetine to improve the quality-of-life interference of CIPN using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity 4 Item version. Exploratory outcomes include i) Determine the difference between the proportion of participants treated with methadone compared to duloxetine that have a 30% and a 50% reduction in average pain intensity; ii) Assess the efficacy of methadone compared to duloxetine to improve the patients' global impression of change (PGIC) using the PGIC questionnaire; iii) Assess the incidence of adverse events with methadone compared to duloxetine using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0, and iv) assess dose tolerance of longer-term methadone use via the Opioid-Escalation Index.

Anticipated Impact: This study will determine if methadone is a viable treatment for CIPN: a very common, distressing, and debilitating condition that otherwise has limited treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old.
2. Estimated life expectancy greater than 12 weeks.
3. Opioid naïve or oral morphine equivalent use <60 mg/day.
4. Greater than grade 1 CIPN based on CTCAE.
5. >3/10 average CIPN-related neuropathic pain lasting ≥3 months beyond chemotherapy completion.
6. A cancer diagnosis.
7. Treatment with one of the following neurotoxic chemotherapies: platinums, taxanes, vinca alkaloids, bortezomib, or thalidomide.

Exclusion Criteria:

1. Other causes of peripheral neuropathy.
2. The following psychiatric illnesses: severe depression, suicidality, bipolar disease or psychotic disorder, alcohol or substance use disorder, DSM V criteria eating disorder.
3. The following medical illnesses: known or suspected mechanical gastrointestinal obstruction or any disease/conditions that affect bowel transit, suspected surgical abdomen, acute or severe asthma, COPD, acute respiratory depression, elevated serum CO2 and cor pulmonale, delirium tremens, convulsive disorders, severe CNS depression such as from cerebrospinal or intracranial pressure and head injury, diarrhea from pseudomembranous colitis, leptomeningeal disease.
4. Liver or renal dysfunction within the last 90 days as defined by MELD-Na score ≥17 and GFR ≤30 ml/min respectively.
5. QTC >499ms within last 90 days.
6. Current pregnancy or lactation.
7. Inability to take oral medications.
8. Positive CAGE and/or Opioid Risk Tool - Revised questionnaire
9. Known allergy or hypersensitivity to opioids, duloxetine, or any ingredient in their formulation.
10. Concomitant use of excluded medications: methadone, other antidepressants (including within 14 days of discontinuing monoamine oxidase inhibitors), thioridazine, potent CYP1A2 inhibitors (such as fluvoxamine and some quinolone antibiotics).
11. Uncontrolled narrow-angle glaucoma.
12. If women of child-bearing potential (i.e. Menstruation within <2 years) are unable or unwilling to use Health Canada approved highly effective methods of contraception (hormonal contraceptives, intrauterine device or system, vasectomy, tubal ligation, or double barrier method), or abstinence during the treatment period.

Note: Any use of prior co-analgesics will be continued (and must have been stable for more than 2 weeks), but the use of new co-analgesics or titration of current co-analgesics will not be permitted during the trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of methadone compared to duloxetine to reduce the reported average pain intensity using the Brief Pain Inventory-Short Form questionnaire. | 5 weeks
  This is a well validated tool that is independently completed by participants. It measures pain intensity and the functional interference caused by pain via four items assessing average, worse, least, and immediate pain intensity in the last 24 hours. Pain intensity is measured using an 11-point numeric rating scale (0=no pain; 10=worst you can imagine). The participant's "average" pain intensity will be the primary end-point; this will be aligned with other clinical trials on chemotherapy-induced peripheral neuropathy (CIPN) and will facilitate comparison across studies.

SECONDARY OUTCOMES:
Efficacy of methadone compared to duloxetine to improve the functional interference of CIPN using the Brief Pain Inventory-Short Form questionnaire. | 5 weeks
  This tool additionally measures seven items assessing the interference of pain on daily activities/function (0=does not interfere; 10=completely interferes), which will be summed to obtain a total interference score out of 70.
Efficacy of methadone compared to duloxetine to improve the quality-of-life interference of CIPN using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity 4 Item version. | 5 weeks
  This is another well validated tool that evaluates quality of life affected by peripheral neuropathy and was, in part, created for clinical trials specifically including CIPN.
  It contains 11 questions ultimately assessing joint pain or muscle cramps, discomfort, numbness or tingling in hands or feet, weakness all over, trouble hearing, tinnitus, trouble buttoning buttons, feeling small shapes when placed in the hand. Items are scored from 0-4 (0=not at all; 4=very much) and summed (total score range=0-44).

OTHER OUTCOMES:
Difference between the proportion of participants treated with methadone compared to duloxetine that have a 30% and a 50% reduction in average pain intensity. | 5 weeks
  This will help differentiate if there are "methadone-responders". This will detect if there is a significant proportion of patients with 30% and 50% pain reduction in the methadone group compared to placebo even if the reduction in average pain intensity is only modest.
Efficacy of methadone compared to duloxetine to improve the Patients' Global Impression of Change (PGIC) using the PGIC questionnaire. | 5 weeks
  This again is a well validated tool designed specifically to assess patients' perception of changes following treatment. It is a 7-point verbal scale with the options "very much improved," "much improved," "minimally improved," "no change," "minimally worsened," "much worsened," and "very much worsened." The PGIC is commonly used in clinical studies involving pain including peripheral neuropathy.
Incidence of adverse events with methadone compared to duloxetine using the National Cancer Institute Common Terminology Criteria for Adverse Events v5.0. | 5 weeks
  This ubiquitous system will be used to classify the severity and incidence of adverse events as reported by participants.
Dose tolerance of longer-term methadone use via the Opioid-Escalation Index (OEI). | 24 weeks
  The OEI will be calculated by determining the difference in methadone total daily dose 12 and 24 weeks after treatment completion. Understanding the OEI for methadone is crucial for managing long-term pain therapy, as it helps minimize the risks of adverse events while ensuring effective pain control.

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Nanaimo Regional Hospital, Nanaimo, British Columbia
  - BC Cancer Surrey, Surrey, British Columbia
  - BC Cancer Vancouver, Vancouver, British Columbia
  - BC Cancer Victoria, Victoria, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belayneh M, Hejazi S, Gagnon B, Hawley P. Methadone to treat chemotherapy-induced peripheral neuropathy (METACIN): study protocol. Pain Manag. 2025 May;15(5):235-243. doi: 10.1080/17581869.2025.2494495. Epub 2025 Apr 28. PMID 40289780